CLINICAL TRIAL: NCT06742138
Title: A Randomized, Multicenter, Double-Blind, Parallel-Controlled, Phase III Clinical Study to Evaluate QL2109/ DARZALEX FASPRO® in Combination With Pomalidomide and Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma Who Have Received at Least One Prior Line of Therapy With Both Lenalidomide and a Proteasome Inhibitor
Brief Title: To Evaluate the Efficacy and Safety of QL2109 and DARZALEX FASPRO® in Multiple Myeloma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QL2109-301
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pomalidomide Plus(+) QL2109 + Dexamethasone (Experimental)
  Interventions: Drug: QL2109; Drug: Pomalidomide; Drug: Dexamethasone
- Pomalidomide + DARZALEX FASPRO® + Dexamethasone (Active Comparator)
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone; Drug: DARZALEX FASPRO®

INTERVENTIONS:
Drug: QL2109 — QL2109 will be given 1800 mg subcutaneously at weekly intervals (QW) for 8 weeks, then every 2 weeks (Q2W) for an additional 16 weeks, then every 4 weeks (Q4W) thereafter. Subjects will receive pre-infusion medications before infusions to mitigate potential IRRs.
  Arms: Pomalidomide Plus(+) QL2109 + Dexamethasone
Drug: Pomalidomide — Intervention Description：Pomalidomide will be administered at full dose of 4 mg orally (PO) on Days 1 through 21 of each 28-day cycle
Drug: Dexamethasone — Dexamethasone will be administered at a dose of 40 mg (20 mg for patients ≥75 years of age) orally, once daily on Days 1, 8, 15, and 22 of each 28-day treatment cycle
Drug: DARZALEX FASPRO® — DARZALEX FASPRO® will be given 1800 mg subcutaneously at weekly intervals (QW) for 8 weeks, then every 2 weeks (Q2W) for an additional 16 weeks, then every 4 weeks (Q4W) thereafter. Subjects will receive pre-infusion medications before infusions to mitigate potential IRRs
  Arms: Pomalidomide + DARZALEX FASPRO® + Dexamethasone

SUMMARY:
This is a randomized, double-blind, multicenter trial，parallel control designed to evaluate treatment with pomalidomide + QL2109 + dexamethasone compared with pomalidomide + DARZALEX FASPRO® + dexamethasone in the participants with relapsed or refractory Multiple Myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least 18 years of age.
* Subject must have measurable disease of MM as defined by the criteria below:Serum M-protein level ≥0.5 g/dL or urine M-protein level ≥200 mg/24 hours; or Light chain multiple myeloma, for subjects without measurable disease in the serum or urine: Serum immunoglobulin free light chain (FLC) ≥10 mg/dL and abnormal serum immunoglobulin kappa lambda FLC ratio.
* Subjects must have received prior antimyeloma treatment. The prior treatment must have included both a PI- and lenalidomide-containing regimens. Subjects who received only 1 line of prior treatment must have demonstrated PD on or within 60 days of completion of the lenalidomide containing regimen (ie, lenalidomide refractory).
* Subjects must have documented evidence of PD based on the investigator's determination of response as defined by the modified IMWG criteria on or after the last regimen.
* Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 2.
* For subjects experiencing toxicities resulting from previous therapy, the toxicities must be resolved or stabilized to ≤Grade 1.
* Any of the following laboratory test results during Screening:

  1. Absolute neutrophil count ≥1.0 × 109/L;
  2. Hemoglobin level ≥75 g/L (≥4.65 mmol/L); (transfusions are not permitted to reach this level);
  3. Platelet count ≥75 × 109/L in subjects in whom <50% of bone marrow nucleated cells are plasma cells and platelet count ≥50 x 109/L in subjects in whom ≥50% of bone marrow nucleated cells are plasma cells;
  4. Alanine aminotransferase (ALT) level ≤2.5 times the upper limit of normal (ULN);Aspartate aminotransferase (AST) level ≤2.5 x ULN;
  5. Total bilirubin level ≤1.5 x ULN, (except for Gilbert Syndrome: direct bilirubin ≤1.5 × ULN);
  6. Creatinine clearance ≥30 mL/min
  7. Serum calcium corrected for albumin ≤14.0 mg/dL (≤3.5 mmol/L), or free ionized calcium ≤ 6.5 mg/dL (≤1.6 mmol/L).

Exclusion Criteria:

* Subject has plasma cell leukemia (>2.0 × 109/L circulating plasma cells by standard differential) or Waldenström's macroglobulinemia or POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes) or amyloidosis.
* History of malignancy (other than MM) within 3 years before the date of randomization (exceptions are squamous and basal cell carcinomas of the skin, carcinoma in situ of the cervix or breast, or other non-invasive lesion that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence within 3 years).
* Clinical signs of meningeal involvement of MM.
* Previous therapy with any anti-CD38 monoclonal antibody.
* Previous exposure to pomalidomide.
* Subject has received antimyeloma treatment within 2 weeks or 5 pharmacokinetic half-lives of the treatment, whichever is longer, before the date of randomization. The only exception is emergency use of a short course of corticosteroids (equivalent of dexamethasone 40 mg/day for a maximum of 4 days) for palliative treatment before Cycle 1, Day 1 (C1D1).
* Previous allogenic stem cell transplant; or autologous stem cell transplantation (ASCT) within 12 weeks before C1D1.
* Subject has had major surgery within 2 weeks before randomization, or has not fully recovered from an earlier surgery, or has surgery planned during the time the subject is expected to participate in the study or within 2 weeks after the last dose of study drug administration.
* Ongoing ≥ Grade 2 peripheral neuropathy.
* Subject had ≥Grade 3 rash during prior therapy.
* Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Very Good Partial Response (VGPR) or Better | from baseline to week 24
  VGPR or better rate was defined as the percentage of participants who achieved VGPR or complete response (CR) (including stringent complete response[sCR]) according to the IMWG criteria during or after the study treatment.

SECONDARY OUTCOMES:
Percentage of Participants With Very Good Partial Response (VGPR) or Better | from baseline to week 12 and week 48
  VGPR or better rate was defined as the percentage of participants who achieved VGPR or complete response (CR) (including stringent complete response[sCR]) according to the IMWG criteria during or after the study treatment.
Overall Response Rate | from baseline to week 24 and week 48
  Overall response rate is defined as the percentage of randomized subjects who achieve a best response of PR or better using modified IMWG criteria as their best overall response
Overall survival at 18 months | from baseline to 18 months
  the probability of being alive 18 months after randomization